CLINICAL TRIAL: NCT02425943
Title: A Prospective, Open-Label, Multicenter Study to Evaluate the Long-Term Safety of Sculptra®Aesthetic in Immuno-Competent Subjects Stratified by Fitzpatrick Skin Type I-VI)
Brief Title: Sculptra Aesthetic Post-Approval Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLI.04.SPR.US10321
Record Dates: First submitted 2015-04-10; First posted 2015-04-24 (Estimated); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Nasolabial Fold Contour Deficiencies; Wrinkles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sculptra Aesthetic (Experimental)
  Interventions: Device: injectable poly-L-lactic acid Sculptra Aesthetic

INTERVENTIONS:
Device: injectable poly-L-lactic acid Sculptra Aesthetic
  Other Names: Sculptra Aesthetic

SUMMARY:
Study is designed to assess the long-term safety of Sculptra Aesthetic in immune-competent subjects as a single regimen for correction of nasolabial fold (NLF) contour deficiencies and other facial wrinkles.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects seeking correction of shallow to deep NLF contour deficiencies.

Exclusion Criteria:

1. Subjects seeking, at entry into the study, correction of other facial wrinkles with Sculptra Aesthetic in the following anatomical sites/lines: horizontal forehead lines, glabellar frown lines, periorbital lines, periauricular lines, upper lip lines, lower lip lines, corner of the mouth lines and/or horizontal neck folds.
2. Subjects that are less than 18 or greater than 75 years of age.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 867 (Actual)
Dates: Start 2015-05-21 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Operations, Study Chair — Galderma R&D
Locations (18):
- United States (18):
  - Galderma Study Site, Birmingham, Alabama
  - Galderma Study Site, Encino, California
  - Galderma Study Site, Hermosa Beach, California
  - Galderma Study Site, San Diego, California
  - Galderma Study Site, Solana Beach, California
  - Galderma Study Site, Aventura, Florida
  - Galderma Study Site, Boca Raton, Florida
  - Galderma Study Site, Coral Gables, Florida
  - Galderma Study Site, Miami, Florida
  - Galderma Study Site, Buffalo Grove, Illinois
  - Galderma Study Site, Hackensack, New Jersey
  - Galderma Study Site, New York, New York
  - Galderma Study Site, White Plains, New York
  - Galderma Study Site, Nashville, Tennessee
  - Galderma Study Site, Austin, Texas
  - Galderma Study Site, Houston, Texas
  - Galderma Study Site, Plano, Texas
  - Galderma Study Site, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at United States from 21 May 2015 to 28 May 2021.
Pre-assignment Details: A total of 867 participants were enrolled and treated in this study.
Groups:
- Fitzpatrick Skin Types I-III: Participants with Fitzpatrick Skin Types I-III received four Sculptra Aesthetic intra-dermal injections with 3-week intervals of multiple 0.1 to 0.2 milliliter (mL) deep dermal injections in a grid pattern, spaced at a distance of approximately 1 centimeter (cm) for up to 9 weeks.
- Fitzpatrick Skin Type IV-VI: Participants with Fitzpatrick Skin Types IV-VI received four Sculptra Aesthetic intra-dermal injections with 3-week intervals of multiple 0.1 to 0.2 mL deep dermal injections in a grid pattern, spaced at a distance of approximately 1 cm for up to 9 weeks.
Period: Overall Study
Arm/Group | Fitzpatrick Skin Types I-III | Fitzpatrick Skin Type IV-VI
Started | 557 | 310
Completed | 421 | 240
Not Completed | 136 | 70
Not completed — Adverse Event | 3 | 1
Not completed — Lost to Follow-up | 59 | 37
Not completed — Protocol Violation | 4 | 1
Not completed — Withdrawal by Subject | 64 | 31
Not completed — Other | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fitzpatrick Skin Type I-III: Participants with Fitzpatrick Skin Type I-III received four Sculptra Aesthetic intra-dermal injections with 3-week intervals of multiple 0.1 to 0.2 mL deep dermal injections in a grid pattern, spaced at a distance of approximately 1 cm for up to 9 weeks.
- Fitzpatrick Skin Type IV-VI: Participants with Fitzpatrick Skin Type IV-VI received four Sculptra Aesthetic intra-dermal injections with 3-week intervals of multiple 0.1 to 0.2 mL deep dermal injections in a grid pattern, spaced at a distance of approximately 1 cm for up to 9 weeks.
- Total: Total of all reporting groups
Arm/Group | Fitzpatrick Skin Type I-III | Fitzpatrick Skin Type IV-VI | Total
Number analyzed (Participants) | 557 | 310 | 867
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (9.25) | 52.6 (9.56) | 54.6 (9.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 524 | 272 | 796
  Male | 33 | 38 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 54 | 123 | 177
  Not Hispanic or Latino | 503 | 187 | 690
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 5 | 5
  Asian | 5 | 9 | 14
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 0 | 88 | 88
  White | 551 | 203 | 754
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 4
Fitzpatrick Classification Skin Type [Count of Participants; unit: Participants] — Skin Type I = White; very fair, red or blonde hair blue eyes; freckles; Always burns, never tans
  Skin Type II = White, fair, red or blond hair; blue, hazel or green eyes; Usually burns, tans with difficulty
  Skin Type III = Cream white; fair with any eye or hair color (common); Sometimes mild burn, gradually tans
  Skin Type IV = Brown; typical Mediterranean Caucasian skin; Rarely burns, tans with ease
  Skin Type V = Dark Brown; mid-eastern skin types; Very rarely burns, tans easily
  Skin Type VI = Black; Never burns, tans very easily
  Participants
    Type I | 32 | 0 | 32
    Type II | 212 | 0 | 212
    Type III | 313 | 0 | 313
    Type IV | 0 | 168 | 168
    Type V | 0 | 96 | 96
    Type VI | 0 | 46 | 46

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Any Injection Site Nodule and/or Papule
Description: Nodules and/or papules are a subset of AEIs that does not include hypertrophic scarring, keloid formation, changes in skin pigmentation at the site of injection compared to adjacent skin, granuloma (confirmed by a biopsy), skin necrosis, hypersensitivity reactions, and unexpected changes in wrinkle contour. Reporting of a nodule or papule was based on size (nodule greater than or equal to [>=] 0.5 (cm); papule less than [<] 0.5 cm). Percentage of participants with any injection site nodule and/or papule were reported.
Time Frame: Up to 5 years
Population: Intent to treat (ITT) Population included all participants who received at least one injection of study drug.
Measure: Number; unit: percentage of participants
Groups:
- Fitzpatrick Skin Types I-III: Participants with Fitzpatrick Skin Types I-III received four Sculptra Aesthetic intra-dermal injections with 3-week intervals of multiple 0.1 to 0.2 mL deep dermal injections in a grid pattern, spaced at a distance of approximately 1 cm for up to 9 weeks.
Arm/Group | Fitzpatrick Skin Types I-III | Fitzpatrick Skin Type IV-VI
Number analyzed (Participants) | 557 | 310
percentage of participants | 30.52 | 24.84

2. Primary Outcome: Percentage of Participants With Any Adverse Events of Interest (AEIs)
Description: AEIs means: "serious or non-serious adverse event that is one of scientific and medical concern specific to the sponsor's product for which ongoing monitoring and rapid communication by the investigator to the sponsor can be appropriate. Examples of AEIs were hypertrophic scarring, keloid formation, hypersensitivity reactions, skin necrosis, unexpected change in wrinkle contour, granuloma, changes in the skin pigmentation at the site of injection compared to adjacent. Percentage of participants with any AEIs (other than injection site nodule and/or papule) were reported.
Time Frame: Up to 5 years
Population: ITT Population included all participants who receive at least one injection of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Fitzpatrick Skin Types I-III | Fitzpatrick Skin Type IV-VI
Number analyzed (Participants) | 557 | 310
Percentage of participants | 30.9 | 25.8

3. Secondary Outcome: Change From Baseline in Nasolabial Folds (NLF) Wrinkle Assessment Score (WAS) at Months 6, 13, and Years 2, 3, 4, and 5
Description: NLF severity was assessed by the evaluating investigator from WAS. WAS was based on a 6-point assessment grade where 0=no wrinkles; 1=just perceptible wrinkle; 2=shallow wrinkle; 3=moderately deep wrinkle; 4=deep wrinkle, well-defined edges; 5=very deep wrinkle, redundant fold. The calculations for average WAS was based on data corresponding to only the nasolabial folds (NLFs) treated at the initial visit, that is., only WAS scores for treated sides was considered. The average WAS was calculated from the individual left and right NLFs scores. If the WAS was only available for one side, then the average WAS was the score for the one side.
Time Frame: Baseline, Months 6,13 and Years 2,3 4,5
Population: ITT Population included all participants who received at least one injection of study drug. "Here, 'overall number of participants analyzed' signifies participants who were evaluable for this outcome measure and "number analyzed" signifies participants who were evaluable for given time points.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Fitzpatrick Skin Type IV-VI: Participants with Fitzpatrick Skin Types IV-VI received four Sculptra Aesthetic intra-dermal injections with 3-week intervals of multiple 0.1 to 0.2 milliliter (mL) deep dermal injections in a grid pattern, spaced at a distance of approximately 1 cm for up to 9 weeks.
Arm/Group | Fitzpatrick Skin Types I-III | Fitzpatrick Skin Type IV-VI
Number analyzed (Participants) | 504 | 271
Score on a scale
  At Month 6 | -1.73 (0.826) | -1.82 (0.847)
  At Month 13: number analyzed (Participants) | 495 | 271
  At Month 13 | -1.74 (0.785) | -1.70 (0.801)
  At Year 2: number analyzed (Participants) | 467 | 252
  At Year 2 | -1.60 (0.833) | -1.63 (0.836)
  At Year 3: number analyzed (Participants) | 169 | 67
  At Year 3 | -1.16 (0.908) | -1.25 (0.937)
  At Year 4: number analyzed (Participants) | 417 | 240
  At Year 4 | -0.80 (0.927) | -0.95 (0.916)
  At Year 5: number analyzed (Participants) | 418 | 239
  At Year 5 | -0.47 (0.883) | -0.62 (0.994)

4. Secondary Outcome: Change From Baseline in Cheek Folds Wrinkle Assessment Score (WAS) at Months 6, 13, and Years 2, 3, 4, and 5
Description: The WAS is a validated photograph-based outcome instrument that is designed specifically for quantifying facial folds. The physician assessed the left side and the right side of the participant's face using the 5-point scale where scoring of wrinkle severity (grades 0-5, with 0 representing no wrinkles and 5 representing very deep wrinkles, redundant fold) was based on visual live assessment by the investigator at defined timepoints. Higher scores mean a worse outcome.
Time Frame: Baseline, Months 6,13 and Years 2,3 4,5
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Fitzpatrick Skin Types I-III | Fitzpatrick Skin Type IV-VI
Number analyzed (Participants) | 128 | 29
Score on a scale
  At Month 6 | -1.54 (0.835) | -1.88 (0.988)
  At Month 13: number analyzed (Participants) | 126 | 28
  At Month 13 | -1.49 (0.924) | -1.96 (0.849)
  At Year 2: number analyzed (Participants) | 117 | 27
  At Year 2 | -1.47 (0.935) | -1.89 (0.801)
  At Year 3: number analyzed (Participants) | 110 | 25
  At Year 3 | -1.30 (1.038) | -1.74 (0.818)
  At Year 4: number analyzed (Participants) | 100 | 25
  At Year 4 | -0.93 (1.179) | -1.38 (1.044)
  At Year 5: number analyzed (Participants) | 99 | 24
  At Year 5 | -0.62 (1.255) | -1.08 (1.283)

5. Secondary Outcome: Change From Baseline in Marionette Lines Wrinkle Assessment Score (WAS) at Months 6, 13, and Years 2, 3, 4, and 5
Description: Marionette Lines severity was assessed by the evaluating investigator from WAS. WAS was based on a 6-point assessment grade where 0=no wrinkles; 1=just perceptible wrinkle; 2=shallow wrinkle; 3=moderately deep wrinkle; 4=deep wrinkle, well-defined edges; 5=very deep wrinkle, redundant fold. The calculations for average WAS was based on data corresponding to only the nasolabial folds (NLFs) treated at the initial visit, that is., only WAS scores for treated sides was considered. The average WAS was calculated from the individual left and right NLFs scores. If the WAS was only available for one side, then the average WAS was the score for the one side.
Time Frame: Baseline, Months 6,13 and Years 2,3 4,5
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Fitzpatrick Skin Types I-III | Fitzpatrick Skin Type IV-VI
Number analyzed (Participants) | 313 | 116
Score on a scale
  At Month 6 | -1.72 (0.831) | -1.87 (0.798)
  At Month 13: number analyzed (Participants) | 311 | 115
  At Month 13 | -1.65 (0.866) | -1.76 (0.825)
  At Year 2: number analyzed (Participants) | 292 | 109
  At Year 2 | -1.52 (0.904) | -1.59 (0.858)
  At Year 3: number analyzed (Participants) | 275 | 105
  At Year 3 | -1.13 (1.023) | -1.24 (1.003)
  At Year 4: number analyzed (Participants) | 262 | 102
  At Year 4 | -0.77 (1.077) | -0.93 (0.989)
  At Year 5: number analyzed (Participants) | 257 | 101
  At Year 5 | -0.41 (1.110) | -0.50 (0.945)

6. Secondary Outcome: Change From Baseline in Chin Crease Wrinkle Assessment Score (WAS) at Months 6, 13, and Years 2, 3, 4, and 5
Description: Chin Crease severity was assessed by the evaluating investigator from WAS. WAS was based on a 6-point assessment grade where 0=no wrinkles; 1=just perceptible wrinkle; 2=shallow wrinkle; 3=moderately deep wrinkle; 4=deep wrinkle, well-defined edges; 5=very deep wrinkle, redundant fold. The calculations for average WAS was based on data corresponding to only the nasolabial folds (NLFs) treated at the initial visit, that is., only WAS scores for treated sides was considered. The average WAS was calculated from the individual left and right NLFs scores. If the WAS was only available for one side, then the average WAS was the score for the one side.
Time Frame: Baseline, Months 6,13 and Years 2,3 4,5
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Fitzpatrick Skin Types I-III | Fitzpatrick Skin Type IV-VI
Number analyzed (Participants) | 200 | 79
Score on a scale
  At Month 6 | -1.54 (0.945) | -1.72 (0.861)
  At Month 13: number analyzed (Participants) | 197 | 76
  At Month 13 | -1.46 (0.992) | -1.71 (0.921)
  At Year 2: number analyzed (Participants) | 183 | 72
  At Year 2 | -1.37 (1.029) | -1.61 (0.987)
  At Year 3: number analyzed (Participants) | 169 | 67
  At Year 3 | -0.99 (1.066) | -1.22 (1.027)
  At Year 4: number analyzed (Participants) | 162 | 65
  At Year 4 | -0.75 (1.075) | -0.86 (1.014)
  At Year 5: number analyzed (Participants) | 160 | 65
  At Year 5 | -0.40 (1.172) | -0.49 (1.048)

7. Secondary Outcome: Percentage of Participants Improved Versus Not Improved on Investigator Assessment of Facial Appearance Using Global Assessment Scale
Description: Efficacy was assessed by overall facial improvement assessed live by the Investigator assessment of facial appearance including the Global Aesthetic Improvement Scale (GAIS). The Global Aesthetic Improvement Scale is a subjective test. The investigator independently describes the degree of improvement in facial appearance. Possible scores were + 3: Much improved, +2: Moderately improved, +1: Slightly improved, 0: No change, -1: Slightly worse, -2: Moderately worse, -3: Much worse. 'Not Improved' included participants with scores of 0, -1, -2, and -3 and 'Improved' included participants with scores of 3, 2, and 1. Higher the GAIS value, the greater the improvement.
Time Frame: At 6,13 months, 2, 3, 4 and 5 years
Population: ITT Population included all participants who receive at least one injection of study drug. "Here, 'Overall number of participants analyzed' signifies participants who were evaluable for this outcome measure and here "number analyzed" signifies participants who were evaluable for this outcome measure for given time points.
Measure: Number; unit: percentage of participants
Arm/Group | Fitzpatrick Skin Types I-III | Fitzpatrick Skin Type IV-VI
Number analyzed (Participants) | 557 | 310
percentage of participants
  Month 6 : Improved | 99.4 | 99.6
  Month 6 : Not Improved | 0.6 | 0.4
  Month 13 : Improved | 99.2 | 99.6
  Month 13 : Not Improved | 0.8 | 0.4
  Year 2 : Improved | 96.6 | 96.0
  Year 2 : Not Improved | 3.4 | 4.0
  Year 3 : Improved | 90.6 | 92.3
  Year 3 : Not Improved | 9.4 | 7.7
  Year 4 : Improved | 80.6 | 82.9
  Year 4 : Not Improved | 19.4 | 17.1
  Year 5 : Improved | 69.6 | 67.5
  Year 5 : Not Improved | 30.4 | 32.5

8. Secondary Outcome: Percentage of Participants Improved Versus Not Improved on Participant Assessment of Facial Appearance Using Global Assessment Scale
Description: Efficacy was assessed by overall facial improvement assessed live by the participants assessment of facial appearance including the GAIS. The GAIS is a subjective test. The participant independently describes the degree of improvement in facial appearance. Possible scores were + 3: Much improved, +2: Moderately improved, +1: Slightly improved, 0: No change, -1: Slightly worse, -2: Moderately worse, -3: Much worse. 'Not Improved' included participants with scores of 0, -1, -2, and -3 and 'Improved' included participants with scores of 3, 2, and 1. Higher the GAIS value, the greater the improvement (Range 0 to 3).
Time Frame: At 6,13 months, 2, 3, 4 and 5 years
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Fitzpatrick Skin Types I-III | Fitzpatrick Skin Type IV-VI
Number analyzed (Participants) | 506 | 273
percentage of participants
  At Month 6 : Improved | 97.2 | 97.8
  At Month 6 : Not Improved | 2.8 | 2.2
  At Month 13 : Improved: number analyzed (Participants) | 496 | 271
  At Month 13 : Improved | 97.4 | 97.4
  At Month 13 : Not Improved: number analyzed (Participants) | 496 | 271
  At Month 13 : Not Improved | 2.6 | 2.6
  At Year 2 : Improved: number analyzed (Participants) | 468 | 252
  At Year 2 : Improved | 91.0 | 92.9
  At Year 2: Not Improved: number analyzed (Participants) | 506 | 252
  At Year 2: Not Improved | 9.0 | 7.1
  At Year 3 : Improved: number analyzed (Participants) | 445 | 249
  At Year 3 : Improved | 85.6 | 88.0
  At Year 3: Not Improved: number analyzed (Participants) | 445 | 249
  At Year 3: Not Improved | 14.4 | 12.0
  At Year 4 : Improved: number analyzed (Participants) | 418 | 241
  At Year 4 : Improved | 73.0 | 76.8
  At Year 4 : Not Improved: number analyzed (Participants) | 418 | 241
  At Year 4 : Not Improved | 27.0 | 23.2
  At Year 5 : Improved: number analyzed (Participants) | 421 | 240
  At Year 5 : Improved | 66.3 | 66.3
  At Year 5: Not Improved: number analyzed (Participants) | 421 | 240
  At Year 5: Not Improved | 33.7 | 33.8

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: ITT Population included all participants who received at least one injection of study drug.
Arm/Group | Fitzpatrick Skin Types I-III | Fitzpatrick Skin Type IV-VI
All-Cause Mortality (participants affected / at risk) | 3/557 | 1/310
Serious Adverse Events (participants affected / at risk) | 39/557 | 11/310
Other Adverse Events (participants affected / at risk) | 315/557 | 150/310
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fitzpatrick Skin Types I-III (N=557) | Fitzpatrick Skin Type IV-VI (N=310)
Granuloma (Congenital, familial and genetic disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Slipping rib syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Diverticulitis (Infections and infestations) | 2 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Corona virus infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Death (General disorders) | 2 | 1
Chest pain (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0
Nerve injury (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Cerebellar haemorrhage (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Pancreas divisum (Congenital, familial and genetic disorders) | 0 | 1
Retinal artery occlusion (Eye disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Granuloma skin (Skin and subcutaneous tissue disorders) | 1 | 0
Knee operation (Surgical and medical procedures) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Multiple sclerosis (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fitzpatrick Skin Types I-III (N=557) | Fitzpatrick Skin Type IV-VI (N=310)
Implant site nodule (General disorders) | 95 | 43
Implant site papules (General disorders) | 101 | 42
Nasopharyngitis (Infections and infestations) | 20 | 5
Sinusitis (Infections and infestations) | 20 | 5
Bronchitis (Infections and infestations) | 13 | 5
Influenza (Infections and infestations) | 7 | 7
Acne (Skin and subcutaneous tissue disorders) | 9 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 3
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 14 | 3
Hypertension (Vascular disorders) | 19 | 3
Hypothyroidism (Endocrine disorders) | 12 | 3
Urinary tract infection (Infections and infestations) | 9 | 1
Corona virus infection (General disorders) | 6 | 3
Upper respiratory tract infection (General disorders) | 7 | 2
Oral herpes (Infections and infestations) | 2 | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 6 | 3
Dermatitis contact (Skin and subcutaneous tissue disorders) | 6 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Osteoporosis (Musculoskeletal and connective tissue disorders) | 7 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 4
Meniscus injury (Injury, poisoning and procedural complications) | 6 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Depression (Psychiatric disorders) | 7 | 1
Seasonal allergy (Immune system disorders) | 4 | 3
Implant site pain (General disorders) | 9 | 4
Implant site discolouration (General disorders) | 1 | 5
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-04-24): https://cdn.clinicaltrials.gov/large-docs/43/NCT02425943/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT02425943/SAP_001.pdf